CLINICAL TRIAL: NCT04634721
Title: Transversus Abdominis Plan Block Applied in Laparoscopic Cholecystectomies Effective By Which Method: Ultrasound or Laparoscopic?
Brief Title: Transversus Abdominis Plan Block, Ultrasound or Laparoscopic?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Mehmet sahap, Principal Investigator, Ankara City Hospital Bilkent
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Ultrasound or Laparoscopic TAP
Record Dates: First submitted 2020-11-01; First posted 2020-11-18 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Bupivacaine; Anesthetics, Local; Anesthetics; Peripheral Nervous System Agents
Keywords: TAP block; laparoscopy; laparoscopic cholecystectomy
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Laparoscopic TAP block (Active Comparator): Laparoscopic assisted TAP block will be done by surgeon intra-operatively
  Interventions: Drug: bupivacaine
- Ultrasaund TAP block (Active Comparator): injecting bupivacaine in transversus abdominis plane to block the somatic nerves
  Interventions: Drug: bupivacaine
- no TAP block (No Intervention): no TAP block would be done

INTERVENTIONS:
Drug: bupivacaine — In one arm the TAP infiltration will contain 10 mL of 0.25 % bupivacaine injected . This will then be repeated on the contralateral side.
  Arms: Laparoscopic TAP block; Ultrasaund TAP block

SUMMARY:
Abdominal wall blocks are frequently used as part of multimodal analgesia for pain control after abdominal surgery. There are studies using the Transversus Abdominis Plane Block for postoperative pain control in laparoscopic cholecystectomies.

In this study, the investigators aimed to compare the advantages of these two methods by applying the Transversus Abdominis Plan Block for postoperative pain control after laparoscopic cholecystectomy with the help of postoperative USG and laparoscopy during surgery.In this study, the investigators aimed to compare the advantages of these two methods by applying the Transversus Abdominis Plan Block for postoperative pain control after laparoscopic cholecystectomy with the help of postoperative USG and LAPAROSCOPY during surgery.

DETAILED DESCRIPTION:
A total of 60 patients aged 18-65, ASA 1-2-3, who will undergo elective laparoscopic cholecystectomy in our hospital, will be included in the study. Patients will be randomly divided into 3 groups with ultrasound (USG) guided (GROUP 1: USG) , Laparoscopic application (GROUP 2: LAP) and GROUP 3 :No-TAP blok Each group consists of 20 evil people. Written consent will be obtained by explaining the procedure to be performed before the operation to the patients. The Transversus Abdominis Plan Block will be applied to the patients by a blind anesthesiologist according to their group. The block to be made by the anesthesiologist who will apply the block procedure will be given in a closed envelope.

ELIGIBILITY:
Inclusion Criteria:

* ASA I,II,III
* Patients 18-65
* laparoscopic cholecystectomy

Exclusion Criteria:

* ASA III higher
* history of pain relief medication dependence
* history of substance abuse
* end stage chronic kidney disease
* advanced liver disease
* history of chronic pain -history of taking opioids or neuropathic agents regularly prior to surgery-
* BMI of 50 or over
* skin infections at the site of TAP block injection or port sites.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
Mean postoperative static and dynamic numeric rating scale (NRS) at 24 hours | 24 hours
  o compare the mean NRS at 0hr, 1hr, 2 hrs. 6 hrs. 12 hrs. and 24hrs. post-operatively between three groups Numeric rating scale for pain,(0=no pain, 1-3= mild pain, 4-6 moderate pain, 7-10 severe pain.)

SECONDARY OUTCOMES:
Post operative nausea or vomiting | 24 hours
  instances of nausea or vomiting in the post operative period will be recorded

OTHER OUTCOMES:
Total opioid usage | 24 hours
  amount of opioids used in perioperative period will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Şehir Hastanesi, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No